CLINICAL TRIAL: NCT04301713
Title: Multifactorial Study of the Relationship Between the Conditions of Life and the Incidence of Risk of Falling, From the Nursing Perspective, in Elderly Adults of the Community
Brief Title: Multifactorial Study of the Relationship Between the Conditions of Life and the Incidence of Risk of Falling
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Prof. Dr. Eduardo J Fernández Rodríguez, Principal Investigator, University of Salamanca
Other Study IDs: 0000281
Record Dates: First submitted 2020-02-04; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Nursing Caries; Old Age; Debility; Aging Disorder
Keywords: older adult; scale, test; risk of falls; life conditions; nursing role
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of rik of falls — An evaluation of the risk of falls will be carried out in the elderly in the province of Salamanca. This will attempt to identify the risk of falling as well as to be able to establish protocols for action of a preventive and rehabilitative nature.

SUMMARY:
HYPOTHESIS:

The incidence of risk of falls is related to the living conditions of elderly people in the community.

OBJECTIVES:

• To study the relationship between living conditions and the incidence of risk of falls in older adults in the community.

SPECIFIC OBJECTIVES:

* Describe the socio-characteristics of the elderly group in the community.
* Identify the pathologies or health problems that they present.
* Evaluate their functional and dependency degree.
* Evaluate the risk of falls that each person may have.
* Identify the risk factors involved in falls.
* Analyze the prevalence of falls that they present.

STUDY DESIGN:

Descriptive and analytical-statistical study. Administration of the Barthel Index. Administration of the Downton fall risk assessment scale and the Falls Efficacy Scale-International (FES-I).

Administration of the Tinetti assessment tool and the Short Physical Performance Battery (SPPB).

Evaluation of socio-demographic characteristics, clinical and functional assessment, consumption of drugs, as well as characteristics of the falls of each elderly person in the community.

The protocol has been authorized by the Ethics Committee of the Salamanca health area to make the project possible.

DETAILED DESCRIPTION:
HYPOTHESIS:

The incidence of risk of falls is related to the living conditions of elderly people in the community.

OBJECTIVES:

• To study the relationship between living conditions and the incidence of risk of falls in older adults in the community.

SPECIFIC OBJECTIVES:

* Describe the socio-characteristics of the elderly group in the community.
* Identify the pathologies or health problems that they present.
* Evaluate their functional and dependency degree.
* Evaluate the risk of falls that each person may have.
* Identify the risk factors involved in falls.
* Analyze the prevalence of falls that they present.

STUDY DESIGN:

Descriptive and analytical-statistical study. Administration of the Barthel Index. Administration of the Downton fall risk assessment scale and the Falls Efficacy Scale-International (FES-I).

Administration of the Tinetti assessment tool and the Short Physical Performance Battery (SPPB).

Evaluation of socio-demographic characteristics, clinical and functional assessment, consumption of drugs, as well as characteristics of the falls of each elderly person in the community.

The protocol has been authorized by the Ethics Committee of the Salamanca health area to make the project possible.

Detailed Description: OBJECTIVES:

To study the relationship between living conditions and the incidence of risk of falls in the elderly group in the community.

SPECIFIC OBJECTIVES:

* Describe the socio-characteristics of the elderly group in the community.
* Identify the pathologies or health problems that they present.
* Evaluate their functional and dependency degree.
* Evaluate the risk of falls that each person may have.
* Identify the risk factors involved in falls.
* Analyze the prevalence of falls that they present.

STUDY DESIGN:

Observational, cross-sectional study. Administration of the Barthel Index. Administration of the Downton fall risk assessment scale and the Falls Efficacy Scale-International (FES-I).

Administration of the Tinetti assessment tool and the Short Physical Performance Battery (SPPB).

Evaluation of socio-demographic characteristics, clinical and functional assessment, consumption of drugs, as well as characteristics of the falls of each elderly person in the community.

Analyze statistically the results obtained and interpret them. The study was carried out over three years. This research study was approved by the Bioethics Committee of the University of Salamanca.

SITE - SAMPLE SELECTION:

The study will include men and women, aged 75 or older, citizens of Salamanca city, who voluntarily participate in the study, during the years 2018-2020, and are attached to the National Health System.

SAMPLE SIZE:

The sample size of the study will be calculated through the estimate of the population of inhabitants of the city of Salamanca in the last year.

The sample technique is intentional. Participants who have met the previously established inclusion criteria and who did not present any exclusion criteria are recruited, as long as they expressed their consent in the participation of the study, voluntarily and altruistically, when they are asked by the nurse. If so, they will be cited later to conduct a separate personal interview.

INDEPENDENT VARIABLES:

• Demographic data of the subject: age, sex, marital status, profession, lifestyle (lives alone: yes/no and housework help: yes/no), weight, height, body mass index, pathological antecedents, pharmacological treatment and history of falls.

DEPENDENT VARIABLES:

• Habitual physical activity, characteristics of falls, risk of falls and fear of falling.

DESCRIPTION OF THE INTERVENTION: Process description

1. Subjects interested in participating in the study will receive a Participant Information Sheet, explaining the objectives and procedures of the research study. It also refers to the principles of non-maleficence, autonomy and participation and voluntary withdrawal, data protection and confidentiality.
2. All the participants included in the study will be identified with a unique number (the selection number) to guarantee anonymity. The code that identifies them will appear in each source of the study.
3. Socio-demographic data of the subjects, pathological history, falls and habitual medication are collected.

   The subjects are evaluated on the risk of falls, the basic activities of daily life and walking and balance, fragility and fear of falling, through the administration of the scales: the Barthel Index, the Downton fall risk assessment scale, the Falls Efficacy Scale-International (FES-I) and the Tinetti assessment tool and the Short Physical Performance Battery (SPPB).
4. The final phase consists on analyze statistically the results obtained and interpret them.

ETHICAL-LEGAL ASPECTS OF THE PROJECT: The protocol has been authorized by the Ethics Committee of the Salamanca health area to make the project possible

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 75 or older.
2. Citizens of Salamanca city, in Spain.
3. People who are attached to the National Health System.
4. Potential candidates who express consent to participate in the study.

Exclusion Criteria:

1. People bedridden for illness in the last three months.
2. Terminal patients or with diagnosis of severe cognitive impairment.
3. Living in nursing homes or homes for the elderly.
4. Potential candidates who do not express consent to participate in the study.

Withdrawal Criteria:

1. Participants who decide to leave the study in any of its phases.
2. People who leave the National Health System in Salamanca to go to another community.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: People over 75 years of the province of Salamanca who are not institutionalized.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Risk of falls | 26/5000 January 2017 - up to 24 weeks
  Psychometric characteristics of the scale, the following criteria will be analyzed:
  * Reproducibility: reliability study (homogeneity of measurements).
  * Validity: content (the items of the instrument adequately represent the construct that it intends to measure) and criteria (degree of similarity in scale scores compared to a standard or reference standard).

CONTACTS AND LOCATIONS:
Locations (1):
- Irene Escosura Alegre, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
A specific database will be created to which any external researcher can access after contacting by email with the PI (mail: ire.escosura@usal.es)
Supporting Information: Study Protocol, SAP, ICF, CSR

DOCUMENTS (1):
  • Informed Consent Form (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT04301713/ICF_000.pdf